CLINICAL TRIAL: NCT00830011
Title: Cognitive Behavioral Therapy for Painful Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Robert Kerns, PhD; Chief, Psychology Service (PI), VA Connecticut Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RK0029; DF03-35
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Neuropathy
Keywords: diabetes; neuropathy; chronic pain; Cognitive behavioral therapy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (Active Comparator): Medical care including medication for neuropathic pain
  Interventions: Other: standard medical care
- CBT (Active Comparator)
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — Ten sessions of manualized CBT delivered by a PhD level psychologist
  Arms: CBT
Other: standard medical care — any care recommended by physician for treatment of diabetic neuropathy including medication.
  Arms: standard care

SUMMARY:
The primary objective of this study is to evaluate the usefulness of cognitive behavioral therapy (CBT) for the management of painful diabetic neuropathy. Participants will be randomly assigned to one of two treatment conditions: CBT plus standard medical care or standard medical care alone. CBT will be offered in ten, ninety-minute group sessions and will be provided by a psychologist with experience in the management of both diabetes and chronic pain. CBT will involve teaching and encouraging practice of adaptive pain coping skills such as relaxation skills, activity pacing, and positive self-statements, among others. This study will allow us to determine which treatment is superior in terms of improvements in pain management, functioning and overall quality of life.

DETAILED DESCRIPTION:
Research Design: A randomized mixed factorial controlled design will be employed in which CBT plus standard pharmaceutical care (CBT/SC) is compared to a standard pharmaceutical care (SC) treatment condition. Participants will be randomized in equal numbers to the two conditions. Repeated assessments of key outcome domains will occur at pretreatment/baseline and at 12, 24 and 36 weeks following baseline.

Methodology: Study participants will be evaluated pre-treatment (baseline), 12 weeks post-baseline (post-treatment) and at 24 and 36 weeks post-baseline (follow-up). Baseline assessment will include a neurological examination with a nerve conduction study to confirm the diagnosis of diabetic neuropathy. The primary outcome measure will be pain intensity. Secondary outcome measures will be pain quality, pain-related disability, physical and emotional functioning. Measures of treatment feasibility will also be examined. Participants receiving CBT will attend 10 weekly, group treatment sessions of 90 minutes. A target sample size of approximately 120 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* daily lower extremity pain or discomfort (burning, tingling or other parasthesias) for at least 3 months
* documented trial of at least one medication for neuropathic pain
* pain of at least 4 on a 0-10 numeric rating scale

Exclusion Criteria:

* acute medical condition, substance abuse, or psychiatric condition that would impair ability to participate
* dementia (MMSE score of 23 or lower)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity score (NRS) | post treatment and follow-up (24 and 36 weeks)

SECONDARY OUTCOMES:
pain-related disability (MPI) and emotional functioning | post treatment and followup (24 and 36 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kerns, PhD, Principal Investigator — VA Connecticut Healthcare System

REFERENCES:
- [Derived] Higgins DM, Heapy AA, Buta E, LaChappelle KM, Serowik KL, Czlapinski R, Kerns RD. A randomized controlled trial of cognitive behavioral therapy compared with diabetes education for diabetic peripheral neuropathic pain. J Health Psychol. 2022 Mar;27(3):649-662. doi: 10.1177/1359105320962262. Epub 2020 Oct 19. PMID 33070667
- See also: American Diabetes Association — http://www.diabetes.org